CLINICAL TRIAL: NCT05062642
Title: Validation of a Predictive Rule for the Diagnosis of Viral Meningitis in Adult Emergency Departments
Acronym: Adult-BMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2020/S02/20
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-09

CONDITIONS: Meningitis
Keywords: BMS score; Meningitis
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Meningitis is the development of an inflammatory reaction in the meningeal space, most often of infectious origin. Many pathogens can cause meningitis, the severity of which varies greatly. Patients presenting with a febrile meningeal syndrome are most often managed in the emergency room, where the challenge for physicians is to quickly differentiate bacterial and viral meningitis.

Viral meningitis is the most common, with enterovirus meningitis having a classically excellent prognosis. Bacterial meningitis is less frequent but more serious.The current public health objective is to save antibiotics.

Investigator hypothesizes that the BMS score can be used to exclude bacterial meningitis in the emergency department in an adult European population of patients with suspected bacterial meningitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the Adult Emergency Department of CH Le Mans,CHU Angers, CHU Nantes or Beaujon Hospital.
* Over 18 years old
* Having had a lumbar puncture during their stay in the Adult Emergency Department
* Having had a diagnosis of meningitis defined as a pleocytosis ≥ 5leukocytes/mm3 after correction with CSF red blood cells at a standardized ratio of 500/1.

Exclusion Criteria:

* Antibiotic therapy within 72 hours of inclusion
* Immunosuppression from any cause
* Presence of petechiae or purpura
* History of recent neurosurgery or head trauma
* Other associated bacterial infection
* Inability to collect information for the BMS score calculation or primary endpoint (e.g., transfer to another facility)
* Minor or adult patient under guardianship or protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be extracted from the population having consulted the Adult Emergency Departments of the Le Mans Hospital, the Angers and Nantes University Hospitals and the Beaujon University Hospital between January 1, 2009 and December 31, 2020 and for whom a lumbar puncture will have been performed for suspected meningitis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-08-26 (Estimated); Study Completion 2022-08-26 (Estimated)

PRIMARY OUTCOMES:
External validation of the BMS score in a European adult population to exclude bacterial meningitis | 1 month after inclusion
  Validation was measured by comparaison between BMS score and the diagnosis retained from the data collected in the file

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France